CLINICAL TRIAL: NCT02671695
Title: Effect of Spirulina Compared to Amlodipine on Cardiac Iron Overload in Children With Beta Thalassemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Professor Mohamed Elshanshory, head of pediatric hematology and oncology unit, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22/03/15
Record Dates: First submitted 2016-01-30; First posted 2016-02-02 (Estimated); Last update posted 2018-07-12 (Actual); Status verified 2017-10

CONDITIONS: Beta Thalassemia Major
MeSH Terms: conditions — beta-Thalassemia | interventions — Amlodipine

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): chelation therapy plus Spirulina capsules (500 mg) in a dose of 250 mg/kg/day orally for 3 months
  Interventions: Drug: Spirulina
- Group 2 (Experimental): chelation therapy plus Amlodipine in a dose of 5 mg/day orally for 3 months
  Interventions: Drug: Amlodipine

INTERVENTIONS:
Drug: Spirulina — Spirulina capsules (500 mg) in a dose of 250 mg/kg/day orally for 3 months
  Arms: Group 1
Drug: Amlodipine — Amlodipine in a dose of 5 mg/day orally for 3 months
  Arms: Group 2

SUMMARY:
the aim of this study is to evaluate the effect of Spirulina compared to Amlodipine on cardiac iron overload and cardiac functions in multi-transfused children with beta thalassemia major

DETAILED DESCRIPTION:
the aim of this study is to evaluate the effect of Spirulina compared to Amlodipine on cardiac iron overload using magnetic resonance imaging and cardiac functions in multi-transfused children with beta thalassemia major

ELIGIBILITY:
Inclusion Criteria:

* patients on regular blood transfusions.
* iron overload with no perspective of changing the chelation therapy in the following three months

Exclusion Criteria:

* formal contraindication to magnetic resonance examinations
* implantable cardiac device
* advanced cardiomyopathy or conduction block
* other types of hemolytic anemias

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2015-04; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
cardiac iron concentration by magnetic resonance imaging | 3 months

SECONDARY OUTCOMES:
cardiac troponin 1 | 3 months
N-terminal pro-brain natriuretic peptide | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Sahar M El-Haggar, MD, Principal Investigator — assisstant professor of clinical pharmacy- Faculty of Pharmacy- Tanta University
Locations (1):
- Faculty of Medicine- Tanta University, Tanta, Gharbia Governorate, Egypt

REFERENCES:
- [Derived] Padhani ZA, Gangwani MK, Sadaf A, Hasan B, Colan S, Alvi N, Das JK. Calcium channel blockers for preventing cardiomyopathy due to iron overload in people with transfusion-dependent beta thalassaemia. Cochrane Database Syst Rev. 2023 Nov 17;11(11):CD011626. doi: 10.1002/14651858.CD011626.pub3. PMID 37975597